CLINICAL TRIAL: NCT01739465
Title: A Randomized Controlled Trial Comparing Endoscopic Biliary Radiofrequency Ablation With Photodynamic Therapy for Inoperable Cholangiocarcinoma
Brief Title: Comparison of Endoscopic Radiofrequency Ablation Versus Photodynamic Therapy for Inoperable Cholangiocarcinoma
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Huihong Liang, Associated Professor, Guangzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RFA2012
Record Dates: First submitted 2012-11-29; First posted 2012-12-03 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Cholangiocarcinoma
Keywords: Cholangiocarcinoma; Pathologic; Digestive System; Neoplasms; Neoplasms by Site; Digestive System Diseases; Bile Duct Diseases; Biliary Tract Diseases; Pathological Conditions; Constriction; Adenocarcinoma; Carcinoma
MeSH Terms: conditions — Cholangiocarcinoma; Neoplasms; Neoplasms by Site; Digestive System Diseases; Bile Duct Diseases; Biliary Tract Diseases; Constriction, Pathologic; Adenocarcinoma; Carcinoma | interventions — Photochemotherapy

ARMS (3):
- Self expanding metallic stent （SEMS ）placement only (Active Comparator): Endoscopic retrograde cholangiopancreatography (ERCP) or percutaneous transhepatic cholangiography (PTC) would be performed to confirm the position and length of the biliary malignant. A self expanding metallic stent (SEMS) would be placed to bypass the site of narrowing
  Interventions: Procedure: Self expanding metallic stent (SEMS)
- Endoscopic radiofrequency ablation plus SEMS (Experimental): Endoscopic retrograde cholangiopancreatography (ERCP) or percutaneous transhepatic cholangiography (PTC) would be performed to confirm the position and length of the biliary malignant. The radiofrequency ablation (RFA) catheter (EMcision, London, United Kingdom) would be placed under fluoroscopic guidance across the biliary stricture. Radiofrequency energy will be delivered to the malignant site. After that,A self expanding metallic stent (SEMS) would be placed to bypass the site of narrowing
  Interventions: Procedure: Self expanding metallic stent (SEMS); Procedure: Endoscopic radiofrequency ablation (ERFA)
- Photodynamic therapy plus SEMS (Experimental): Photofrin is injected 3 days prior to laser activation of the agent.Endoscopic retrograde cholangiopancreatography (ERCP) or percutaneous transhepatic cholangiography (PTC) will be carried out to determine the length and positon of the biliary malignant. Delivery Fiber used along with the laser system to activate the photosensitizing agent and induce tumor tissue necrosis. A self expanding metallic stent (SEMS) will be placed the site of biliary narrowing
  Interventions: Procedure: Self expanding metallic stent (SEMS); Procedure: Photodynamic therapy (PDT)

INTERVENTIONS:
Procedure: Self expanding metallic stent (SEMS) — Self expanding metallic stent
Procedure: Endoscopic radiofrequency ablation (ERFA) — Endoscopic radiofrequency ablation
  Arms: Endoscopic radiofrequency ablation plus SEMS
Procedure: Photodynamic therapy (PDT) — Photodynamic therapy
  Arms: Photodynamic therapy plus SEMS

SUMMARY:
The purpose of this study is to compare endoscopic radiofrequency ablation with photodynamic therapy for inoperable cholangiocarcinoma

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Pathologically or radiologically confirmed biliary malignant
* Inoperability by staging

Exclusion Criteria:

* Cholangiocarcinoma with widespread metastasis
* Coagulopathy (INR > 2.0 or prothrombin time > 100 sec or platelet count < 50,000)
* Prior SEMS placement
* Pregnancy
* Eastern Cooperative Oncology Group (ECOG) performance status ≥ 3 )
* Life expectancy < 3months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2012-11; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
stent patency | 6 months

SECONDARY OUTCOMES:
overall survival rate | 3 years

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - The Second Hospital of Guangzhou Medical College, Guangzhou, Guangdong
  - The second hospital of Guangzhou Medical college, Guangzhou, Guangdong